CLINICAL TRIAL: NCT06742411
Title: A Phase Ib/II Clinical Trial of the XELOX Regimen Combined With Sintilimab and Hyperbaric Oxygen Therapy for the Treatment of Advanced or Metastatic Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: XELOX Combined With Sintilimab and HBO for Advanced or Metastatic GC/GEJC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Liu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCH20242269
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Gastric (Stomach) Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XELOX+Sintilimab+HBOT (Experimental): Patients will receive the XELOX regimen, consisting of oxaliplatin (130 mg/m² IV on Day 1) and capecitabine (1000 mg/m² orally twice daily for 14 days, repeated every 3 weeks), combined with sintilimab (200 mg IV on Day 1 every 3 weeks) and hyperbaric oxygen therapy (HBOT) administered alongside the XELOX regimen. Treatment will be administered for 4 to 6 cycles.
  Following the initial treatment phase, patients will be evaluated for response. If disease progression is observed, patients will exit the study and receive subsequent treatments as deemed appropriate. For patients with stable disease or a response to therapy, maintenance treatment with capecitabine and sintilimab will continue until the occurrence of a study endpoint or other specified criteria.
  Interventions: Drug: XELOX+Sintilimab+HBOT

INTERVENTIONS:
Drug: XELOX+Sintilimab+HBOT — Patients will receive the XELOX regimen, consisting of oxaliplatin (130 mg/m² IV on Day 1) and capecitabine (1000 mg/m² orally twice daily for 14 days, repeated every 3 weeks), combined with sintilimab (200 mg IV on Day 1 every 3 weeks) and hyperbaric oxygen therapy (HBOT) administered alongside the XELOX regimen. Treatment will be administered for 4 to 6 cycles.
  Following the initial treatment phase, patients will be evaluated for response. If disease progression is observed, patients will exit the study and receive subsequent treatments as deemed appropriate. For patients with stable disease or a response to therapy, maintenance treatment with capecitabine and sintilimab will continue until the occurrence of a study endpoint or other specified criteria.

SUMMARY:
This study investigates the efficacy and safety of XELOX chemotherapy combined with sintilimab and hyperbaric oxygen therapy (HBOT) as a first-line treatment for patients with Advanced or Metastatic gastric and gastroesophageal junction adenocarcinoma. The trial comprises two phases: a phase Ib study to determine the optimal HBOT regimen and assess safety and tolerability, followed by a phase II study to evaluate the overall response rate (ORR). Secondary outcomes include progression-free survival (PFS), disease control rate (DCR), 2-year disease-free survival (DFS), 2-year overall survival (OS), safety, and quality of life. This study aims to provide a novel approach for enhancing therapeutic efficacy and improving patient outcomes by leveraging HBOT to address tumor hypoxia and augment the effects of chemotherapy and immune checkpoint inhibitors.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase Ib/II clinical trial designed to evaluate the safety and efficacy of the XELOX regimen combined with sintilimab and hyperbaric oxygen therapy (HBOT) in patients with Advanced or Metastatic gastric and gastroesophageal junction adenocarcinoma.

In the phase Ib portion, 9 patients will be enrolled to identify the optimal HBOT protocol and assess the safety and tolerability of the combined treatment. The dose and schedule of HBOT will be refined based on observed safety data and adverse events.

In the phase II portion, approximately 48 patients will be enrolled to further evaluate the efficacy of the XELOX plus sintilimab and HBOT combination. Patients will receive treatment in 3-week cycles, with HBOT administered alongside chemotherapy and immunotherapy. The primary endpoint of the phase II study is the overall response rate (ORR) assessed per RECIST 1.1 criteria.Secondary endpoints include progression-free survival (PFS), disease control rate (DCR), 2-year disease-free survival (DFS), 2-year overall survival (OS), safety profile, and patient-reported outcomes related to quality of life. Exploratory endpoints will focus on biomarker analysis and the role of HBOT in modulating tumor hypoxia.This study aims to explore whether HBOT can enhance the efficacy of chemotherapy and immunotherapy by addressing tumor hypoxia, a known factor contributing to therapy resistance in gastric and gastroesophageal junction cancers. The findings from this trial may provide insights into a novel multimodal treatment strategy for improving patient outcomes in advanced disease settings.

ELIGIBILITY:
Inclusion criteria:

1.Diagnosis: Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (including signet ring cell carcinoma, mucinous adenocarcinoma, and hepatoid adenocarcinoma).

2.Disease status: The presence of metastatic disease, attributable to either recurrence or distant dissemination, was established through a combination of radiologic or surgical assessments.

3.Survival Expectancy: Predicted to live more than 3 months. 4.Age: 18-75 years. 5.Prior treatments:

1. There are no previous antitumor treatments (chemotherapy, radiotherapy, targeted therapy, immunotherapy, interventional therapy, etc.).
2. If patients previously received adjuvant or neoadjuvant therapy, the last treatment must have been completed at least 6 months before randomization, with no recurrence or disease progression during treatment.
3. Palliative radiotherapy is allowed if it is completed at least 2 weeks before the first study treatment.
4. The use of prior anti-tumor traditional Chinese medicine is allowed if it is discontinued at least 2 weeks before randomization.

6.Performance Status: ECOG PS ≤1. 7.Assessable lesion: At least one measurable lesion per the RECIST 1.1 criteria.

8.Pathological samples: Patients whose archived or fresh pathological tissue was obtained within 6 months before signing informed consent, which was sufficient for PD-L1 testing with obtainable results, were included.

9.Organ function:

1. Hematology (no transfusion or G-CSF use within 14 days before screening):

   Hemoglobin ≥90 g/L. Absolute neutrophil count (ANC) ≥1.5×10⁹/L. Platelet count ≥75×10⁹/L.
2. Biochemistry (no albumin use within 14 days before screening):

Albumin ≥28 g/L. Total bilirubin ≤1.5×ULN. AST and ALT levels were ≤3×ULN (≤5×ULN if liver metastasis was present). creatinine ≤1.5×ULN. (3)Coagulation: INR or PT ≤1.5×ULN. APTT ≤1.5×ULN. 10.Systemic treatment history: No systemic treatment (including adjuvant/neoadjuvant) was given within the past 6 months after sample collection for randomization.

11.Toxicity: Prior antitumor treatment or surgery-related acute toxic reactions were resolved to grade 0-1 per NCI CTCAE v5.0 or to levels specified by the inclusion/exclusion criteria.

12.Contraception: Strict contraception measures. 13.Consent and Compliance: Signed informed consent, willing and able to comply with study visits, treatments, lab tests, and procedures.

Exclusion criteria:

1. HER2 status: HER2-positive (HER2 3+ or 2+ & FISH+).
2. Tumor type: Nonadenocarcinoma gastric cancers, including squamous cell carcinoma, undifferentiated carcinoma, or mixed histological types.
3. CNS Metastasis: Uncontrolled or symptomatic active CNS metastasis (e.g., clinical symptoms, brain edema, spinal cord compression, carcinomatous meningitis, soft meningeal disease, or progressive growth).
4. Fluid accumulation: Uncontrolled pleural effusion or ascites treated with drainage within 14 days before randomization; symptomatic or moderate to large pericardial effusion.
5. Weight loss: Weight loss >20% within 2 months before randomization.
6. Recent treatments:

(1)Major surgery within 28 days before randomization (diagnostic biopsies and PICC placement allowed).

(2)Immunosuppressive drugs should be used within 7 days before randomization, excluding nasal/inhaled corticosteroids or physiological-dose systemic steroids (≤10 mg/day prednisone or equivalent).

(3)Live attenuated vaccines were administered within 28 days before randomization, during the study, or within 60 days after treatment ended.

(4)Antitumor treatments were administered within 28 days before randomization (chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy, or tumor embolization).

7.Other Malignancies: Patients were diagnosed with any other malignancy within 3 years before study entry, except for localized and cured basal cell carcinoma, squamous or superficial bladder carcinoma, cervical carcinoma in situ, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma.

8.Autoimmune Diseases: Any active, known, or suspected autoimmune disease. Stable conditions not requiring systemic immunosuppression are allowed (e.g., type I diabetes; hypothyroid diabetes managed with hormone replacement; and skin diseases not needing systemic treatment, such as vitiligo, psoriasis, and alopecia).

9.Neurological/Psychiatric Conditions: Uncontrolled epilepsy, congenital spherocytosis, claustrophobia, or angle-closure glaucoma.

10.Immune therapy history: Prior treatment with anti-PD-1/PD-L1 antibodies, anti-CTLA-4 antibodies, or other T-cell costimulation/checkpoint pathway drugs.

11.Bleeding/thrombosis events: significant bleeding symptoms or tendencies within 3 months before randomization; gastrointestinal perforation or fistula within 6 months; thrombotic events (e.g., stroke, deep vein thrombosis, pulmonary embolism) within 6 months.

12.Major Vascular Disease: Major vascular disease within 6 months before study treatment (e.g., aortic aneurysm needing surgery or recent peripheral arterial thrombosis).

13.Wounds and fractures: Severe, unhealed, or open wounds; active ulcers; or untreated fractures.

14.Neuropathy: Peripheral neuropathy >Grade 1. 15.Intestinal Obstruction: History of intestinal obstruction or related symptoms within 6 months before study treatment. Patients treated surgically to resolve incomplete obstructions at initial diagnosis may be included.

16.Systemic diseases: Interstitial lung disease, noninfectious inflammation, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, acute pneumonia).

17.Drug Allergies: Patients with known severe allergic reactions to the study drugs or any monoclonal antibodies.

18.HIV/AIDS: HIV infection or known AIDS. 19.Hepatitis: Untreated active hepatitis B (HBV-DNA ≥500 IU/ml), hepatitis C (HCV-RNA above the detection limit), or coinfection with HBV and HCV.

20.Cardiac conditions: Myocardial infarction, severe/unstable angina, NYHA Class II or higher heart failure, significant arrhythmias, or congestive heart failure within 6 months before randomization.

21.Hypertension: Poorly controlled hypertension despite treatment (systolic BP >140 mmHg or diastolic BP >90 mmHg).

22.Infections and Fever: Systemic antibiotic use ≥7 days within 4 weeks before randomization or unexplained fever >38.5°C during screening/before the first dose (tumor-related fever allowed on the basis of the investigator's judgment).

23.Transplant history: Known history of allogeneic organ or hematopoietic stem cell transplantation.

24.Other Clinical Trials: Participation in any other drug clinical trial within 4 weeks before randomization or within 5 half-lives of the last study drug.

25.Substance Abuse: History of psychiatric drug abuse or drug addiction. 26.Other Severe Conditions: Any other serious physical or mental illness, abnormal lab tests increasing study risk or interfering with results, or deemed unsuitable by the investigator.

27.The pulmonary conditions were as follows: treated pneumothorax, severe emphysema, or pulmonary bullae.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | ORR will be assessed after 4 to 6 cycles of treatment (approximately 12 to 18 weeks). Evaluation will include imaging performed at baseline and at the end of the treatment cycles to determine the tumor response.
  The primary outcome measure is the overall response rate (ORR), defined as the proportion of patients achieving a complete response (CR) or partial response (PR) as assessed by RECIST 1.1 criteria. ORR will be evaluated based on imaging and clinical assessments conducted during the study.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment to the first disease progression or death, assessed up to approximately 24 months.
  Progression-free survival (PFS) is defined as the time from the start of treatment to the first documented disease progression, as assessed by RECIST 1.1 criteria, or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | After 4-6 cycles of treatment (approximately 12-18 weeks).
  Disease control rate (DCR) is defined as the proportion of patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) as assessed by RECIST 1.1 criteria.
Downstaging Rate | After 4-6 cycles of treatment (approximately 12-18 weeks).
  Downstaging rate is defined as the proportion of patients whose tumors are successfully reduced in stage, enabling resection or improved therapeutic options, as determined by imaging and clinical evaluations.
2-Year Disease-Free Survival (DFS) | From the start of treatment to 2 years post-treatment.
  Two-year disease-free survival (DFS) is defined as the percentage of patients who remain free of disease recurrence after achieving disease control or response to treatment within the study period.
2-Year Overall Survival (OS) | From the start of treatment to 2 years post-treatment.
  Two-year overall survival (OS) is defined as the percentage of patients who are still alive 2 years after initiating treatment, regardless of disease progression.
Adverse Events | From the start of treatment to the end of the study (up to approximately 24 months).
  Safety will be assessed based on the incidence, nature, and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) graded according to the NCI-CTCAE v5.0.
Quality of Life (QoL) | Baseline, every 3 weeks during treatment, and every 12 weeks post-treatment, up to 24 months.
  Quality of life (QoL) will be evaluated using validated patient-reported outcome measures, such as the EORTC QLQ-C30 questionnaire, to assess the physical, emotional, and functional well-being of patients during and after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li W, Zhang P, Cheng M, Wei J, Xu M, Li D, Song S, Liu M, Huang C, Zhu L. XELOX combined with sintilimab and hyperbaric oxygen therapy for advanced or metastatic gastric/gastroesophageal junction adenocarcinoma: study protocol for a prospective, single-arm, phase Ib/II clinical trial. Front Immunol. 2026 Jan 12;16:1672725. doi: 10.3389/fimmu.2025.1672725. eCollection 2025. PMID 41601634